CLINICAL TRIAL: NCT05860712
Title: Evaluation Of Antimicrobial Potency Of A Novel Cinnamon Extract Irrigant Versus Sodium Hypochlorite Irrigant Following Pulpectomy Of Primary Teeth . (A Randomized Clinical Trial)
Brief Title: Evaluation of Antimicrobial, Post Operative Pain of Cinnamon Extract Versus Sodium Hypochlorite Irrigant Following Pulpectomy of Primary Teeth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amany Hossam, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17279
Record Dates: First submitted 2023-05-06; First posted 2023-05-16 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Irreversible Pulpitis; Caries,Dental
Keywords: antimicrobial and post operative pain evaluation
MeSH Terms: conditions — Dental Caries | interventions — Therapeutic Irrigation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium hypochlorite Irrigation (Active Comparator): standardized pulpectomy procedure will be performed using a large sterile round end bur in a high-speed handpiece with copious irrigation, and a sharp spoon excavator will remove pulpal tissues to the orifice level , the working lengths of root canals were estimated by apex locator and Cleaning and shaping of the root canals was done by rotary files .The pre - irrigation sample were collected after debridement of the radicular pulp tissues by a sterile paper point ,then Second microbial sample : The canals were irrigated with Sodium hypochlorite Irrigation (group A) .All the microbiological culturing procedures were carried out in the Microbiology and Immunology Department , the plates were examined and the colonies were directly counted using colony forming unit .
  Interventions: Other: Irrigation
- Cinnamon extract Irrigation (Sham Comparator): standardized pulpectomy procedure will be performed using a large sterile round end bur in a high-speed handpiece with copious irrigation, and a sharp spoon excavator will remove pulpal tissues to the orifice level , the working lengths of root canals were estimated by apex locator and Cleaning and shaping of the root canals was done by rotary files .The pre - irrigation sample were collected after debridement of the radicular pulp tissues by a sterile paper point ,then Second microbial sample : The canals were irrigated with cinnamon Irrigation (group B) . All the microbiological culturing procedures were carried out in the Microbiology and Immunology Department , the plates were examined and the colonies were directly counted using colony forming unit .
  Interventions: Other: Irrigation

INTERVENTIONS:
Other: Irrigation — Cinnamon to be prepared were mixed with 50% ethanol and this suspension was placed on the magnetic stirrer for 4 hours.Whitman's filter paper was used to obtain the filtrate which was then dried to obtain the extract. The extract was dried to evaporate the solvent to prevent the influence of extracting agent (ethanol) on the final extract. Cinnamon extract was obtained using cinnamon bark which was pulverized into medium coarse granules. The extracting agent and the procedure to obtain the final extract.These extracts were stored in dark coloured bottles at 4 degree Celsius until use.

SUMMARY:
The aim of the study is to evaluate effectiveness of cinnamon extract versus sodium hypochlorite as root canal irrigant for in pulpectomy of primary teeth in reduction of bacterial count .

DETAILED DESCRIPTION:
Preservation of primary teeth with non-vital pulp is a major problem in pediatric dentistry, as it is a poly-microbial and dominated by obligatory anaerobic bacteria. Regarding these case preferable treatment modality is pulpectomy . The objective of pulpectomy is complete removal of necrotic and irreversibly infected pulp of an affected tooth but due to limited ability of mechanical preparation to eliminate entrapped micro-organisms in the canal space owing to the tortuous and complex nature of the root canal system .Thus, the use of antimicrobial agents has been recommended as an adjunct to mechanical instrumentation in deciduous teeth . Due to potential side effects, safety concerns of synthetic drugs and cytotoxic reactions of commercial intra canal irrigants and their limited ability to eliminate bacteria from dentinal tubules . Finding the best irrigating solution for endodontic therapy in primary and permanent teeth is still a working progress .There is a growing interest in using sustainable products of natural origin as an alternative to commercially available industrial ones .Cinnamon , which has gained popularity in recent time due its antibacterial , antifungal , anti-inflammatory & antiseptic activity . It has shown effectiveness against S. mutans and E. fecalis organisms . It is also known to show a wide spectrum of action on gram positive and gram negative bacteria .

ELIGIBILITY:
Inclusion Criteria:

* Children:

  1. Aged 4 to 8, in good general health, and medically free.
  2. Cooperative patients who will comply to dental treatment .
  3. Parents provided with written informed consent.
  4. No previous history of antibiotics administration or last dose was taken from at least 2 weeks.
* Teeth:

  1. Carious primary molars with irreversible pulpitis.
  2. Presence of localized swelling ,sinus and pain on percussion which indicate non vital pulp .
  3. Presence of periapical and furcation radiolucency .
  4. In periapical radiograph teeth have no more than 1/3 of root resorption.

Exclusion Criteria:

* Children:

  1. Children with medical, physical, or mental conditions.
  2. Severly Uncooperative children .
* Teeth:

  1. Primary molars with any congenital anomalies.
  2. Teeth with un-restorable crowns .
  3. Root resorbtion more than half of the root.

     -

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-11-22 (Estimated)

PRIMARY OUTCOMES:
Change in bacterial count. | Day 1
  Quantitative.(Colony Forming Unit ) take sample by paper point before and after irrigation by control of interventional

SECONDARY OUTCOMES:
post operative pain evaluation | 6,12,24,48,72 hour
  four point facial pain intensity scoring system

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt